#### RESEARCH SUBJECT CONSENT FORM

TITLE: A Randomized, Controlled, Masked (Reading Center)

Prospective Study of the Effectiveness and Safety of the Ocular Therapeutix Dextenza (dexamethasone Ophthalmic insert) 0.4 mg for the treatment of post-operative inflammation and pain in patients who have undergone

PhotoREfractive Keratectomy (PRK)-

**PROTOCOL NO.:** The RESTORE Study

ASPIRE® Protocol #20201216

SPONSOR: John P. Berdahl, MD
INVESTIGATOR: John P. Berdahl, MD
SITE(S): Vance Thompson Vision

3101 W 57th St

Sioux Falls, South Dakota 57108

**United States** 

SUB-INVESTIGATOR: Mitch Ibach, OD

Study-Related

**Phone Number(s):** 605-361-3937

605-361-3937 (24 hours)

### **RESEARCH CONSENT SUMMARY**

You are being asked for your consent to take part in a research study. This document provides a concise summary of this research. It describes the key information that we believe most people need to decide whether to take part in this research. Later sections of this document will provide all relevant details.

#### What should I know about this research?

- Someone will explain this research to you.
- Taking part in this research is voluntary. Whether you take part is up to you.
- If you don't take part, it won't be held against you.
- You can take part now and later drop out, and it won't be held against you
- If you don't understand, ask questions.
- Ask all the guestions you want before you decide.

# How long will I be in this research?

We expect that your taking part in this research will last approximately 12-14 weeks.

# Why is this research being done?

The purpose of this research is to evaluate the efficacy and safety of Dextenza for the treatment of postoperative pain and inflammation following Photorefractive Keratectomy (PRK) surgery compared to a standard steroid drop regimen. The use of DEXTENZA (dexamethasone ophthalmic insert) 0.4 mg in this study is considered investigational.

## What happens to me if I agree to take part in this research?

If you decide to take part in this research study, the general procedures include 6 visits, including one surgery day and 5 office visits, as well as 1 phone call survey. The study will have 2 groups; one group of 10 eyes that will receive Dextenza and one group of 10 eyes that will receive topical steroid drops. Each participant will have one eye in each group. You will also receive topical antibiotic drops to be used in both eyes for one week.

# Could being in this research hurt me?

The risks associated with participation in this clinical research study are expected to be similar to other therapeutic corticosteroid topical drop options for the treatment of postoperative pain and inflammation following PRK surgery and may include bacterial infections, viral infections, fungal infections, increased intraocular pressure, and glaucoma. Previous studies in adults have shown that treatment with Dextenza is safe and well tolerated in a similar patient population that underwent ophthalmic surgery.

## Will being in this research benefit me?

The most important benefits that you <u>may</u> expect from taking part in this research is reduction of pain and inflammation post-surgery.

# What other choices do I have besides taking part in this research?

Instead of being in this research, your choices may include a current standard of care topical corticosteroid ophthalmic drop regimen or Dextenza. Please discuss with your doctor other alternatives that may be available to you.

#### **DETAILED RESEARCH CONSENT**

You are being invited to take part in a research study because you are scheduled to have PRK surgery in both your eyes. A person who takes part in a research study is called a research subject, or research participant.

#### What should I know about this research?

- Someone will explain this research to you.
- This form sums up that explanation.
- Taking part in this research is voluntary. Whether you take part is up to you.
- You can choose not to take part. There will be no penalty or loss of benefits to which you are otherwise entitled.
- You can agree to take part and later change your mind. There will be no penalty or loss of benefits to which you are otherwise entitled.

- If you don't understand, ask questions.
- Ask all the questions you want before you decide.

## Why is this research being done?

The purpose of this research is to evaluate the efficacy and safety of Dextenza for the treatment of postoperative pain and inflammation following PRK surgery. This is a prospective, single-center, open-label clinical trial; it is being conducted only here at your doctor's office, and both you and your physician will know the treatment type and dosage of the study medication. Each eye will receive a different steroid therapy after the PRK surgery.

The study drug, Dextenza, is approved by the FDA for the treatment of pain and inflammation following ophthalmic surgery. Dextenza is an intracanalicular insert containing 0.4mg dexamethasone steroid designed to elute preservative-free drug over 30 days. The insert removes the need for topical administration of dexamethasone (or other similar steroid) eye drops in that eye following surgery.

The other eye will receive topical dexamethasone or similar steroid eye drops.

About 20 subjects will take part in this research.

## How long will I be in this research?

We expect that your taking part in this research will last approximately 12-14 weeks.

# What happens to me if I agree to take part in this research?

During the study, the following procedures will be done. Some of these exams will happen more than once while you are in the study.

- **Medical/Surgical History:** You will also be asked questions about your overall health, past diseases, and surgeries.
- **Concomitant Medications:** You will be asked questions about the medications, vitamins, or other supplements you take.
- **Demographics:** You will be asked questions such as your date of birth, race, and ethnic background.
- Adverse Events: You will be asked question to find out whether you are having any changes in health or side effects during the study.
- **Numerical Rating Scale (NRS Pain Scale):** You will be asked to rate your pain from 0 (no pain) to 10 (most pain).
- **SPEED Questionnaire:** You will be asked questions about your dry eye symptoms.
- **COMTOL Questionnaire:** You will be asked questions about your personal experience and satisfaction with the study insert.
- **Urine Pregnancy Test:** If you are a woman able to have children, you must have a pregnancy test by giving a urine sample.

- The study doctor or staff will tell you if the pregnancy test results are positive.
   The results of the pregnancy testing must be negative for you to stay in the study.
- Best Corrected Visual Acuity: Your vision will be measured using an eye chart.
- **Slit-Lamp Biomicroscopy:** The study doctor will look into the front of your eye using a machine that has a bright light.
- **IOP** (Intraocular Pressure): You will have drops put in your eyes to numb them. Once your eyes are numb, the pressure inside of your eyes will be measured by using a machine that gently touches the surface of your eyes.
- Dilated Fundus Examination: The study doctor will put dilating drops in your eyes, once your eyes are dilated, the doctor will look at the back of your eye with a bright light.
- Pentacam: A special light beam will be used to take a picture of the inside of you eve.
- Insertion of Dextenza: The study drug is a small insert that is placed in the punctum, a natural opening in the eye lid. The study doctor will first apply anesthetic drops to the eye to numb the eye. The study doctor will then place a small probe into the punctum to open the punctum to allow for the insert. The insert will then be placed into the punctum with forceps, which are like tweezers. Normal saline drops will then be applied to your eye.
- Application of 1% prednisolone acetate: You will be required to insert the drops 4 times a day for a week and then 2 drops a day for an additional week in the eye that did not receive the Dextenza insert.

#### **Screening Visit**

Before you do anything in this study, you will be asked to sign and date this consent form. A copy of the signed and dated consent form will be given to you to take home. At this visit, the following procedures and tests will be done:

- Inclusion/exclusion
- Demographics
- Medical History and Concurrent Illnesses
- Concomitant Medications
- Randomization
- Uncorrected Distance visual acuity as measured by ETDRS chart at 4m
- Manifest Refraction
- Best-corrected visual acuity as measured by ETDRS chart at 4m
- Corneal haze (via AS-OCT)
- Intraocular pressure
- Corneal Staining
- Slit Lamp Exam
- Ophthalmic Examination (dilated fundus exam)
- Subject reported AEs prior to or after surgery
- Ocular pain assessment
- Modified Speed questionnaire

#### Surgery Day

At this visit, the following procedures and tests will be done for the study:

- Concomitant medications
- Confirm treatment group
- Record any surgical complications
- Subject reported AEs prior to or after surgery
- Intracanalicular dexamethasone insert in one eye
- Prescribe post-operative topical therapy regimen

#### **Post-Operative Day 3**

At this visit, the following procedures and tests will be done:

- Concomitant medications
- Intraocular pressure
- Corneal staining
- Slit lamp exam
- Subject reported AEs prior to or after surgery
- Insert visualization
- Ocular pain assessment

#### **Post-Operative Day 4**

At this visit, the following procedures and tests will be done:

- Concomitant medications
- Intraocular pressure
- Corneal staining
- Slit lamp exam
- Subject reported AEs prior to or after surgery
- Insert visualization
- Ocular pain assessment

#### Phone Call 1: Day 14

During this call, the following procedures will be done:

- Subject reported AEs prior to or after surgery
- Ocular pain assessment

#### **Post-Operative Day 28**

At this visit, the following procedures and tests will be done:

- Concomitant medications
- Uncorrected Distance visual acuity as measured by ETDRS chart at 4m
- Manifest refraction
- Best-corrected visual acuity as measured by ETDRS chart at 4m
- Corneal haze
- Intraocular pressure
- Corneal staining
- Slit lamp exam
- Subject reported AEs prior to or after surgery
- Insert visualization

- Ocular pain assessment
- Modified Speed questionnaire
- Adapted COMTOL Survey

#### **Post-Operative Month 3**

At this visit, the following procedures and tests will be done:

- Concomitant medications
- Uncorrected Distance visual acuity as measured by ETDRS chart at 4m
- Manifest refraction
- Best-corrected visual acuity as measured by ETDRS chart at 4m
- Corneal haze
- Intraocular pressure
- Corneal staining
- Slit lamp exam
- Subject reported AEs prior to or after surgery
- Insert visualization

## What are my responsibilities if I take part in this research?

If you take part in this research, you will be responsible to:

- Follow the instructions you are given.
- Come to the study clinic for all visits with the study doctor or study staff.
- Tell the study doctor or study staff about any changes in your health or the way you feel.
- Tell the study doctor or study staff about any changes in your medications or new medications you may have taken.
- Tell the study doctor or study staff if you want to stop being in the study at any time.

It is important for you to be honest with your study doctor about your medical history and any medicines or supplements you are taking in order to prevent any harm to you in taking part in this study.

# Could being in this research hurt me?

The risks associated with participation in this clinical research study are expected to be similar to other corticosteroid therapeutic options for the treatment of postoperative pain and inflammation following PRK surgery. Side effects from the Dextenza and the topical steroid drops may include:

- bacterial infections.
- viral infections,
- fungal infections,
- increased intraocular pressure,
- pain
- swelling
- redness and

#### • glaucoma.

Previous studies in adults have shown that treatment with Dextenza is safe and well tolerated in an appropriate patient population. The most common non-eye side effect experienced was a headache.

One of the reasons for this study is to learn more about the safety and efficacy of Dextenza for the treatment of postoperative pain and inflammation following PRK surgery. It is important that you tell the study staff about possible complications you experience while participating in the study. Not all risks can be predicted. If you have any health-related problems during your treatment, you should contact the Principal Investigator (John Berdahl, MD) of the study at Vance Thompson Vision, Sioux Falls as soon as possible. It is not possible to predict in advance if any problems will develop, but if they do occur you will be promptly treated. The study protocol also permits your doctor to administer "rescue medication", or a different medication that he/she sees as an option for you in the case that Dextenza is not working for your pain and inflammation. A possible side effect to any of the investigational drugs is an allergic reaction. If you experience any allergic reactions please notify the study doctor.

## Will it cost me money to take part in this research?

There will be no additional cost to you for taking part in this research.

## Will being in this research benefit me?

There have been positive findings with use of the dexamethasone insert in the treatment of postoperative pain and inflammation. You may benefit by having your pain and inflammation reduced, however there is no promise your pain and inflammation will be reduced. Information from this study might help researchers to come up with new tests or medications to help others in the future.

# What other choices do I have besides taking part in this research?

There are other treatments available for postoperative pain and inflammation. Currently, corticosteroid ophthalmic topical drops are used for the treatment of postoperative pain and inflammation in PRK surgery.

You do not need to participate in this study to be treated for your condition. You should discuss your alternatives to participating in this research with the study doctor or study staff. In addition, you may discuss your options with your regular health care provider.

# What happens to the information collected for this research?

Your private information and your medical record will be shared with individuals and organizations that conduct or watch over this research, including:

- The research sponsor
- People who work with the research sponsor
- Government agencies, such as the Food and Drug Administration
- The Institutional Review Board (IRB) that reviewed this research

We may publish the results of this research. However, we will keep your name and other identifying information confidential.

We protect your information from disclosure to others to the extent required by law. We cannot promise complete secrecy.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

Efforts will be made to keep your study-related information confidential. However, there may be circumstances where this information must be released. For example, personal information regarding your participation in this study may be disclosed if required by state law.

Also, your records may be reviewed by the following groups (as applicable to the research):

- Office for Human Research Protections or other federal, state, or international regulatory agencies;
- U.S. Food and Drug Administration;
- The sponsor supporting the study, their agents or study monitors
- The Institutional Review Board (IRB) that reviewed this research

If this study is related to your medical care, your study-related information may be placed in your permanent hospital, clinic, or physician's office records. You may also be asked to sign a separate Health Insurance Portability and Accountability Act (HIPAA) research authorization form if the study involves the use of your protected health information.

# Who can answer my questions about this research?

If you have questions, concerns, or complaints, or think this research has hurt you or made you sick, talk to the research team at the phone number listed above on the first page.

This research is being overseen by an Institutional Review Board ("IRB"). An IRB is a group of people who perform independent review of research studies. You may talk to them at 1-877-366-5414 (toll-free), <a href="mail@aspire-irb.com">email@aspire-irb.com</a> if:

- You have questions, concerns, or complaints that are not being answered by the research team.
- You are not getting answers from the research team.
- You cannot reach the research team.
- You want to talk to someone else about the research.
- You have questions about your rights as a research subject.

# What if I am injured because of taking part in this research?

In the event that you should be injured in the course of a research study, you will be provided with the necessary medical care at Vance Thompson Vision. However, this statement does not mean that either such medical care of hospitalization, if necessary, will be free of charge. Furthermore, we cannot provide you with compensation as a result of any injury. If you are injured as a result of this study, you do not give up your right to pursue a claim through the legal system.

## Can I be removed from this research without my approval?

The study doctor may end your participation in the study without your permission at any time. The Sponsor may also choose to terminate the entire study at any time. Your participation to the study could be terminated for example, if you are unable to follow the study procedures or if medical events occur that could impact your safety, or if too many subjects have been enrolled. If you are withdrawn from the study, you may be asked to have the appropriate medical tests and follow-up to evaluate your health and safety.

# What happens if I agree to be in this research, but I change my mind later?

Participation in this study is voluntary and it is entirely your decision whether or not you take part in this study. If after reading this information and talking with the medical staff you choose not to take part, or if you change your mind after agreeing and signing the consent form, for any reason, your decision will be respected. If you decide not to participate in this study, or end your participation for any reason, you may receive a standard treatment, and no prejudice or bias will be show toward you for routine medical care.

You can stop taking part in this study at any time. If you decide to take part in this study, but later withdraw for any reason, study data collected prior to your withdrawal may still be used.

If you decide to stop being part of the study you should:

- tell the study doctor immediately;
- see the study doctor to be examined

If you withdraw your consent to participate in this study, then no new information will be collected from you with the exception of information for adverse events occurring at the time of your withdrawal.

# Will I be paid for taking part in this research?

You will not receive compensation for your participation in the study. You will receive PRK at no cost to you.

# **Statement of Consent:**

| Your signature documents your consent to take part in this research. | |
|---|---|
| Signature of adult subject capable of consent | Date |
| Signature of person obtaining consent | Date |
| dignature of person obtaining consent | Bate |
| My signature below documents that the information in the consent form and any other written information was accurately explained to, and apparently understood by, the subject, and that consent was freely given by the subject. | |
| Signature of witness to consent process | Date |